CLINICAL TRIAL: NCT06510088
Title: Prognostic Impact of a 3-week Multimodal Prehabilitation Program on Frail Elderly Patients Undergoing Elective Gastric Cancer Surgery
Brief Title: Effects of Multimodal Prehabilitation on Frail Elderly Patients Undergoing Elective Gastric Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Senbin Lin, General Surgery, Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TaizhouHospital
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Elderly; Frail; Gastric Cancer; Prehabilitation
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3-week multimodal prehabilitation program+perioperative care guided by ERAS protocols (Experimental): This program included four components: aerobic and resistance exercises, respiratory training, nutritional counseling with whey protein supplementation, and psychological adjustment.
  Interventions: Procedure: 3-week multimodal prehabilitation program
- perioperative care guided by ERAS protocols (No Intervention): Perioperative care of the control group was based on standardized ERAS recommendations that have been widely implemented to minimize heterogeneity in perioperative care. Typically, participants did not receive any preoperative interventions related to exercise, nutrition, or mental health.

INTERVENTIONS:
Procedure: 3-week multimodal prehabilitation program — This program included four components:
  Aerobic and Resistance Exercises A designated physical therapist supervises the resistance exercises and offers corrective guidance. Training intensity was continuously monitored and fine-tuned based on Borg scale assessments.
  Respiratory Training Respiratory training was conducted using a respiratory trainer. Patients were instructed to engage in respiratory training at least three times daily, with each session lasting 10 minutes.
  Nutrition Intervention Those in the multimodal prehabilitation group received daily whey protein powder to ensure a recommended protein intake of 1.5 g/kg/d. Protein supplements were to be consumed within one hour of exercise to promote muscle synthesis.
  Psychological Intervention Anxiety-coping interventions included relaxation techniques and deep breathing exercises, administered in a one-to-one format by a nurse trained in psychological care.
  Arms: 3-week multimodal prehabilitation program+perioperative care guided by ERAS protocols

SUMMARY:
Research indicates that prehabilitation is effective in optimizing physical status before surgery, although this method may be considered "aggressive" for frail elderly patients. This study aimed to evaluate whether multimodal prehabilitation consisting of preoperative physical therapy, nutritional support, and cognitive exercises decreases postoperative complications and improves functional recovery in frail elderly patients undergoing gastric cancer surgery, in comparison to usual clinical care.

DETAILED DESCRIPTION:
Gastric cancer remains a significant health concern globally, especially among elderly individuals, where it poses a considerable burden due to its aggressive nature and limited therapeutic options. Population aging, a result of demographic transition, presents a critical societal challenge. According to a 2022 report by the World Health Organization (WHO), the median age for gastric cancer diagnosis is 69 years, with patients over 75 years facing heightened risks of morbidity and mortality. Although surgical resection remains the primary treatment for gastric cancer, the proportion of elderly patients undergoing surgery declines with age due to preoperative frailty. Frailty, marked by age-related declines in energy, muscle strength, weight, and activity levels, is common among elderly gastric cancer patients and correlates with poorer surgical outcomes, including higher morbidity and mortality. Therefore, interventions aimed at enhancing the functional status and resilience of frail elderly patients undergoing surgery for gastric cancer are critically important.

Numerous studies have demonstrated that prehabilitation can diminish complications, hospital readmissions, length of hospital stay (LOS), and care dependence by enhancing functional reserve. However, these studies did not differentiate between age groups and frailty status, making it difficult to interpret the relationship between the outcomes and advanced age or frailty. It is hypothesized that patients at higher risk for postoperative complications, such as frail elderly individuals, are more likely to benefit from prehabilitation. Nonetheless, conclusive evidence on multimodal rehabilitation specifically designed for this vulnerable population remains insufficient.

Prehabilitation seeks to optimize patients' preoperative risk factors during the waiting period before surgery. This preoperative phase is a critical time to modify health behaviors to reduce the stress of surgery and enhance the recovery process. Multimodal prehabilitation encompasses various interventions, including physical exercise, nutritional optimization, and psychological support, aiming to bolster physiological reserve in anticipation of the expected adverse effects of surgery and to support the postoperative recovery of functional capacity, particularly in patients with lower preoperative fitness levels. Several studies have demonstrated that prehabilitation can diminish complications, hospital readmissions, LOS, and care dependence by enhancing functional reserve. However, during their research, the patients' age group and frailty status were not differentiated, and the relationship between the results and advanced age/frailty cannot be well interpreted. It is hypothesized that patients at higher risk for postoperative complications, such as frail elderly individuals, are more likely to benefit from prehabilitation. Nonetheless, definitive evidence on multimodal rehabilitation specifically tailored to this vulnerable population is lacking.

Therefore, we implemented a randomized clinical trial to provide evidence regarding the potential advantages of multimodal prehabilitation on the outcomes of frail elderly patients undergoing elective gastric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 65;
2. Patients with a Fried Frailty Index score of 2 or higher;
3. Patients who were scheduled for surgical resection of gastric adenocarcinoma;
4. Patients whose life expectancy was estimated by the surgeon to be greater than six months -

Exclusion Criteria:

Patients were excluded from the study if they:

1. were scheduled for neoadjuvant therapy;
2. had metastatic cancer;
3. were unable to swallow or participate in exercise and fitness assessments due to pre-existing conditions (e.g., orthopedic, neuromuscular, or cardiorespiratory diseases);
4. had low compliance, defined as executing less than 70% of the weekly plan;
5. had incomplete data or were lost to follow-up. -

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 30-day after surgery
  30-day postoperative complications assessed by the Comprehensive Complication Index (CCI); The CCI, a validated index for assessing morbidity and mortality, aggregates all complications using the Clavien-Dindo classification system, resulting in a score from 0 (no complications) to 100 (death)
6-minute walking distance (6MWD) | 30-day after surgery3-month after surgery
  Functional capacity was assessed using the 6-MWD, a reliable measure of exercise tolerance in patients undergoing colorectal surgery, with changes of at least 20 meters deemed clinically significant.

SECONDARY OUTCOMES:
recovery of gastrointestinal function | 30 days after surgery
  recovery of gastrointestinal function
QoL | 3-month after surgery
  QoR-9 scale
physical activity | 3-month after surgery
  Short Form (36) health survey (SF-36)
psychological status | 3-month after surgery
  Hospital Anxiety and Depression scale

CONTACTS AND LOCATIONS:
Overall Officials: Senbin Lin, Principal Investigator — Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University
Locations (1):
- Taizhou Hospital of Zhejiang Province Affiliated to Wenzhou Medical University, Taizhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen J, Hong C, Chen R, Zhou M, Lin S. Prognostic impact of a 3-week multimodal prehabilitation program on frail elderly patients undergoing elective gastric cancer surgery: a randomized trial. BMC Gastroenterol. 2024 Nov 11;24(1):403. doi: 10.1186/s12876-024-03490-7. PMID 39528916